CLINICAL TRIAL: NCT00230412
Title: Study of Heat Shock Proteins as Prognostic Factor of Acute Renal Failure in Children (HSP-Study)
Acronym: HSP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Munich Children's Clinic (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Dennis Ballwieser, LMU Munich
Other Study IDs: HSP-233-05; Projektnummer 233-05
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Kidney Failure, Acute
Keywords: Kidney Failure, Acute; Acute Renal Failure; Kidney Failure; Heat-Shock Proteins; Children
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum and urine.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the investigators' study is to determine whether the production of heat shock proteins has an effect on the development and the outcome of acute renal failure in children.

DETAILED DESCRIPTION:
A prognostic factor for the development of acute renal failure (ANR) in children would be very valuable for therapy regulation. So-called chaperones out of the family of heat shock proteins (HSP) are promising candidates which are involved in the development of ANR as well. This could be a starting point for the development of new therapeutic approaches.

ANR occurs in up to 50 percent of all critical ill patients and has a high rate of morbidity and mortality despite advances in symptomatic therapy. Following severe sepsis, septic shock or other shocks, combined with multiple organ failure, the ANR is an autonomous prognosis worsening factor.

Should the results of our study show a correlation between the production of HSP and the outcome of children with ANR, further studies would be required, to examine the pathophysiological relevance of HSP in ANR. We would then be able to determine a high risk population for ANR. A modulation of ANR therapy might be a result of further studies.

ELIGIBILITY:
Inclusion Criteria:

* Between 0 and 18 years of age.
* Either severe sepsis, shock of any origin or asphyxia.
* Operated patients with operative or post-operative transfusion requirement of at least 0.5 x 80 ml/kg body weight of erythrocyte concentrate.

Exclusion Criteria:

* Existing affection of the kidney.
* Kidney transplantation.
* Missing written consent of the parents or guardian (if applicable).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients on paediatric intensive care units.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2005-10; Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Acute renal failure. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Karl Reiter, Dr. med., Study Chair — Klinikum der Universität München, Kinderklinik und Poliklinik im Dr. von Haunerschen Kinderspital; Judith Glöckner-Pagel, Dr. med., Study Director — Klinikum der Universität München, Kinderklinik und Poliklinik im Dr. von Haunerschen Kinderspital; Dennis A. Ballwieser, cand. med., Principal Investigator — Klinikum der Universität München, Kinderklinik und Poliklinik im Dr. von Haunerschen Kinderspital
Locations (6):
- Germany (6):
  - Klinikum Augsburg, II. Klinik für Kinder und Jugendliche, Augsburg, Bavaria
  - Kinderklinik Memmingen, Memmingen, Bavaria
  - Klinikum der Universität München, Kinderklinik und Poliklinik im Dr. von Haunerschen Kinderspital, Munich, Bavaria
  - Deutsches Herzzentrum München, Munich, Bavaria
  - Klinkum der Barmherzigen Brüder St. Hedwig, Regensburg, Bavaria
  - Kinderklinik Rosenheim, Rosenheim, Bavaria

REFERENCES:
- [Background] Lameire N, Van Biesen W, Vanholder R. Acute renal failure. Lancet. 2005 Jan 29-Feb 4;365(9457):417-30. doi: 10.1016/S0140-6736(05)17831-3. PMID 15680458
- [Background] Schrier RW, Wang W. Acute renal failure and sepsis. N Engl J Med. 2004 Jul 8;351(2):159-69. doi: 10.1056/NEJMra032401. No abstract available. PMID 15247356
- [Background] Thadhani R, Pascual M, Bonventre JV. Acute renal failure. N Engl J Med. 1996 May 30;334(22):1448-60. doi: 10.1056/NEJM199605303342207. No abstract available. PMID 8618585
- [Background] Schiffl H, Lang SM, Fischer R. Daily hemodialysis and the outcome of acute renal failure. N Engl J Med. 2002 Jan 31;346(5):305-10. doi: 10.1056/NEJMoa010877. PMID 11821506
- See also: Dr. von Haunersches Kinderspital München/University of Munich Children's Clinic — http://hauner.klinikum.uni-muenchen.de/
- See also: Universität München/University of Munich — http://www.lmu.de
- See also: City of Memmingen Children's Clinic — http://www.kinderklinik-memmingen.de
- See also: City of Augsburg Clinic — http://www.klinikum-augsburg.de
- See also: City of Rosenheim Clinic — http://www.kliro.de
- See also: The Brothers of Mercy's Hospital at Regensburg — http://www.barmherzige-regensburg.de